CLINICAL TRIAL: NCT05117255
Title: Validating an Autonomous Interactive Internet-Based Delivery of an Empirically Supported Cognitive Behavioral Therapy for Comorbidity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00013960
Record Dates: First submitted 2021-09-14; First posted 2021-11-11 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Generalized Anxiety Disorder; Panic Disorder; Social Anxiety Disorder; Alcohol Use Disorder; Depression
MeSH Terms: conditions — Generalized Anxiety Disorder; Panic Disorder; Phobia, Social; Alcoholism; Depression | interventions — Autogenic Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will not know which study group participants have been assigned to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental: Computer-delivered cognitive behavioral therapy hybrid for comorbidity (Experimental): Four, approximately 60 minute each, computerized therapy sessions delivered on an interactive computerized platform. All participants are undergoing a standard 28 day residential alcohol treatment program.
  Interventions: Behavioral: Negative Emotions and Addiction Tools Program (NEAT)- Cognitive Behavioral Therapy
- Control: Progressive Muscle Relaxation Training (PMRT) (Active Comparator): Four, one-hour computerized segments delivered on an interactive computerized platform teaching Progressive Muscle Relaxation Training (PMRT). All participants are undergoing a standard 28 day residential alcohol treatment program.
  Interventions: Behavioral: Progressive Muscle Relaxation Training (PMRT)
- Treatment as Usual (TAU) (No Intervention): Participants are undergoing a standard 28 day residential alcohol treatment program. No study intervention.

INTERVENTIONS:
Behavioral: Negative Emotions and Addiction Tools Program (NEAT)- Cognitive Behavioral Therapy — The program provides simplified clinical, learning and neuroscience-based education about the vicious cycle in which negative affect serves to motivate drinking, which, in turn, worsens negative affect. Participants also learn how each of three skills (breathing control, cognitive restructuring, problem solving) was designed to disrupt a specific element of the vicious cycle that includes physiological, psychological and behavioral processes.
  Arms: Experimental: Computer-delivered cognitive behavioral therapy hybrid for comorbidity
Behavioral: Progressive Muscle Relaxation Training (PMRT) — PMRT is a standard stress management coping skill that entails tensing and releasing specified muscle groups to obtain deep muscle relaxation.
  Arms: Control: Progressive Muscle Relaxation Training (PMRT)

SUMMARY:
This project is designed to determine if a computer-delivered cognitive-behavioral treatment can improve the otherwise poor alcohol use disorder treatment outcomes for individuals with a co-occurring anxiety disorder. In the past, the investigators showed that this treatment does improve outcomes for these individuals when delivered by a therapist. If the present work shows that the computer-delivered version is also effective, it would provide an inexpensive program with virtually unlimited scalability to enable access to the treatment by many more individuals than is currently the case.

DETAILED DESCRIPTION:
The broad goal of the proposed work is to conduct a randomized controlled trial of a specialized computer-delivered cognitive-behavioral therapy (CBT) to supplement standard alcohol use disorder (AUD) treatment in patients with a co-occurring anxiety disorder ("comorbidity"). Comorbidity is both common in AUD treatment patients (up to 50%) and confers a substantial increase in the risk of a return to drinking in the months following treatment. Because research shows that simply adding a standard psychiatric treatment does not substantially improve the AUD outcomes of comorbid individuals, the investigators developed a CBT-based intervention aimed at disrupting the positive-feedback loop ("vicious cycle"; VC) of mutually aggravating negative affect and drinking behavior/urges (the "VC-CBT"). In an Randomized Controlled Trial (RCT), AUD treatment patients who received the therapist-delivered VC-CBT demonstrated significantly improved alcohol use outcomes as compared to those who received a standard anxiety treatment. Unfortunately, most community-based AUD treatment programs do not have clinical staff with the specialized training and technical expertise needed to deliver the VC-CBT. To help bridge this "research-to-practice" gap, the investigators went on to develop a fully autonomous and interactive computer-delivered version of the VC-CBT and have demonstrated its functionality in AUD patients. Now, the investigators propose to test the clinical efficacy of the computer-delivered VC-CBT, as well as the mechanisms and processes by which it is hypothesized to work. Aim I is a randomized controlled trial comparing the computer-delivered VC-CBT to an intensity-matched computer-delivered active control intervention that focuses on healthy lifestyles. 256 individuals in residential AUD treatment who have a comorbid anxiety disorder will receive either the VC-CBT or the active control intervention to obtain 200 cases that complete a 1-, 4- and 8-month follow-up. The investigators predict the VC-CBT group will demonstrate superior alcohol-related outcomes at follow-up relative to the control group. Aim II evaluates the extent to which the computer-delivered VC-CBT selectively imparts the skills targeted and whether they convey (mediate) the interventions therapeutic effect. This entails a formal series of "causal steps" analyses of the associations of: treatment->skills; skills->outcomes; and, treatment -> outcomes, with vs. without the effect of skills->outcomes statistically controlled. Aim III will test the theoretically-derived prediction that the computer-delivered VC-CBT moderates (i.e., weakens) the association of near real-time negative affect and negative situations with drinking behavior and drinking urges. This will be accomplished by analyzing a series of electronic Ecological Momentary Assessment (EMA) recordings completed in participants' natural environment in each of the 30 days following the conclusion of treatment. The impact of this work would be to provide a scalable and inexpensive means of improving the otherwise poor AUD treatment outcomes of comorbid AUD treatment patients. The work will also provide new scientific knowledge about the mechanisms and processes of change stemming from comorbidity treatment.

ELIGIBILITY:
Inclusion Criteria:

* current (past 30 days) Diagnostic and Statistical Manual of Mental Disorders-IV (DSM-IV) diagnosis of panic disorder with or without agoraphobia (PD/Ag), generalized anxiety disorder (GAD) or social anxiety disorder (SAD)
* receiving treatment primarily for alcohol (vs. drug) dependence
* ability to provide informed consent
* a minimum of an eighth grade English reading level
* status as a residential patient in the Lodging Plus (LP) addiction treatment program
* sufficient time left in their residential LP care to complete the study protocol through the post-treatment assessment

Exclusion Criteria:

* cognitive or medical impairments that prohibit study participation as determined by study PI
* serious suicide risk determined by study PI
* court-ordered treatment. (The exclusion is based on its classification as a "vulnerable" population.)
* Self-reported past participation in a Kushner intervention study while in Lodging Plus

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2022-01-04 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Percent heavy ("binge") days drinking | eight-months following treatment (four-month assessment is primary)
  a ratio expressed as a percent of the days the individual drank 5 (for men) or 4 (for women) or more drinks to the total number of days over the follow-up period in which drinking was possible.
Days to first use | eight-months following treatment (four-month assessment is primary)
  Determined for the entirety of the post treatment time for which the investigators have data up to the 8-month assessment.

SECONDARY OUTCOMES:
Any use of alcohol | eight-months following treatment (four-month assessment is primary)
  Any use of alcohol will be binary (yes/no) indicator of whether any alcohol was consumed.
Percent days drinking | eight-months following treatment (four-month assessment is primary)
  a ratio of the days that alcohol was consumed to the total number of possible drinking days.
Days to first binge | eight-months following treatment (four-month assessment is primary)
  Determined for the entirety of the post treatment time for which the investigators have data up to the 8-month assessment.
Days to first 3 consecutive days of drinking | eight-months following treatment (four-month assessment is primary)
  Determined for the entirety of the post treatment time for which the investigators have data up to the 8-month assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Lodging Plus Program, Fairview Hospital, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No